CLINICAL TRIAL: NCT06033131
Title: Preeclampsia Intervention 4 - A Triple Blind Phase III Randomised Controlled Trial Assessing Metformin to Prolong Gestation in Preterm Preeclampsia
Brief Title: PI4 - A Trial Assessing Metformin to Prolong Gestation in Preterm Preeclampsia
Acronym: PI4
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Lina Bergman (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Sponsor-Investigator, Lina Bergman, Senior consultant, Associate Professor, Sahlgrenska University Hospital
Organization: Sahlgrenska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EU Trial nr: 2022-502707-2-00
Record Dates: First submitted 2023-08-28; First posted 2023-09-13 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; Metformin; Preterm birth; Prolongation; Birth weight; Length of stay in neonatal care
MeSH Terms: conditions — Pre-Eclampsia; Premature Birth; Birth Weight | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin ER (Active Comparator): Metformin ER oral tablet 500 mg three times daily and increased to one gram (two tablets) three times daily as tolerated.
  Interventions: Drug: Metformin ER
- Placebo (Placebo Comparator): 1 placebo tablet three times daily and increased to 2 placebo tablets three times daily as tolerated.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin ER — Metformin ER, one gram three times daily taken orally. Once the participants have been recruited, they will start by taking one 500 mg tablet three times a day. If well tolerated it will be increased day two to a maximum of two tablets three times a day. Treatment will continue until delivery. If there are side effects that are not tolerable, the dose will be decreased and the participant will remain blinded. Each participant will keep a treatment diary and number of tablets taken will be documented by the participant or hospital staff. The study will not alter or interfere with treatment or care routinely given for preterm preeclampsia.
  Other Names: Glucophage SR 500 mg prolonged release tablets
  Arms: Metformin ER
Drug: Placebo — Placebo, two tablets three times daily taken orally. Once the participants have been recruited, they will start by taking one tablet three times a day. If well tolerated it will be increased day two to a maximum of two tablets three times a day. Treatment will continue until delivery. If there are side effects that are not tolerable, the dose will be decreased and the participant will remain blinded. Each participant will keep a treatment diary and number of tablets taken will be documented by the participant or hospital staff. The study will not alter or interfere with treatment or care routinely given for preterm preeclampsia.
  Arms: Placebo

SUMMARY:
Preterm preeclampsia is a severe condition for both the mother and the fetus. Currently, the only treatment available to stop disease progression is termination/delivery of the fetus and placenta. Therefore, preterm preeclampsia carries the highest rates of neonatal morbidity and mortality due to iatrogenic preterm birth. There is evidence suggesting metformin, a drug commonly used to treat diabetes in and outside pregnancy, may be able to counter the pathophysiology of preeclampsia, raising the possibility that it could be used to treat the condition. This multi centre double blind randomised controlled trial aims to investigate if metformin can prolong gestation, lower neonatal length of stay and increase birthweight in a Swedish setting.

DETAILED DESCRIPTION:
Preeclampsia is globally responsible for 60,000 maternal deaths per year, and far greater numbers of fetal losses. Preterm preeclampsia is a severe variant with the highest rates of neonatal morbidity and mortality due to iatrogenic preterm birth (clinicians are forced to deliver the baby preterm for maternal or fetal health reasons).

There is preclinical evidence suggesting metformin, a drug commonly used to treat diabetes in and outside pregnancy, may be able to counter the pathophysiology of preeclampsia, raising the possibility that it could be used to treat the condition.

Previous research from the Preeclampsia Intervention 2 trial (PI2) show that metformin was able to delay delivery in early preterm preeclampsia. Metformin extended release (ER) was associated with a median 7.6-day prolongation of pregnancy (geometric mean ratio (GMR) 1.39 (95% CI 0.99 to 1.96) P=0.057).Trends towards increased birthweight (mean difference 110gm (95%CI -80 to 300), a decreased length of stay at the neonatal intensive care unit (median difference 5.0 days less; GMR 0.86, 95% CI 0.62 to 1.2) and a shorter period of admission in any neonatal ward (median difference 12.0 days less; GMR 0.82, 95% CI 0.57 to 1.18) in the metformin ER group were found. Importantly, while gastrointestinal side effects were common, no serious adverse events related to trial medications were observed.

The PI 2 trial has shown that metformin may be a disease modifying treatment for preterm preeclampsia. The trial is being repeated in a larger scale in the PI3 trial in South Africa to also assess neonatal outcomes. In Sweden, the demographics of the population are different and expectant management of preeclampsia allows for the women to reach 37 weeks of gestation as opposed to 34 weeks of gestation in the PI2 trial. This trial aims to investigate if metformin can prolong gestation, lower neonatal length of stay and increase birthweight in a Swedish setting. Follow up of mothers and children will be carried out two years post partum.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of preeclampsia (defined as hypertension in combination with significant proteinuria (albumin/creatinine ratio >8 mg/mmol, protein/creatinine ratio>30 mg/mmol or >2+ protein on a urinary dipstick) has been made by the attending clinician
* The managing clinicians have made the assessment to proceed with expectant management.
* The subject has given written consent to participate in the study.
* The woman must be 18 years of age or older
* The gestational age is between 22+0 weeks to 33+6 weeks with a viable fetus
* The woman carries a singleton pregnancy

Exclusion Criteria:

* Contraindications to treatment with metformin as outlined in SmPC
* Contraindications for expectant management of preeclampsia such as an immediate indication for delivery according to SFOG guidelines for preeclampsia (https://www.sfog.se/media/338533/pe-riktlinje-230214.pdf).
* Type 1 Diabetes Mellitus
* Current use of metformin
* Known or suspected allergies against metformin
* Reluctance or language difficulties that result in difficulty understanding the meaning of study participation
* Unable to understand the informed consent process
* Previous participation in the study
* Established fetal compromise that necessitates imminent delivery (including planned delivery after 48 hours of corticosteroid treatment). This will be decided by the clinical team before expectant management is offered to the patient.
* Suspicion of a major known fetal anomaly or malformation.
* Renal disease or dysfunction, suggested by a creatinine level greater than or equal to 125 µmol/L or rapidly declining renal function
* Known acute or chronic metabolic acidosis, including diabetic ketoacidosis
* Not suitable for inclusion by the opinion of the investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Pregnancy prolongation | From randomisation to delivery, measured in days and hours, up to 105 days
  Length of pregnancy from diagnosis of preeclampsia to delivery

SECONDARY OUTCOMES:
Time for neonatal care | From birth to discharge from neonatal care, measured in days and hours, up to 126 days
  Time for neonatal care from birth to discharge
Neonatal birth weight | At birth
  Birth wight measured in grams

CONTACTS AND LOCATIONS:
Overall Officials: Lina Bergman, Associate professor, Principal Investigator — Sahlgrenska University Hospital
Locations (9):
- Sweden (9):
  - Falu Lasarett, Falun
  - Sahlgrenska University Hospital, Gothenburg
  - Linköping University Hospital, Linköping
  - Skåne University Hospital, Lund
  - Skåne University Hospital, Malmo
  - Karolinska University Hospital Huddinge, Stockholm
  - Karolinska University Hospital Solna, Stockholm
  - Danderyd Hospital, Stockholm
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
We plan to share data with similar ongoing or planned trials in South Africa and The Netherlands.

REFERENCES:
- [Background] Chappell LC, Cluver CA, Kingdom J, Tong S. Pre-eclampsia. Lancet. 2021 Jul 24;398(10297):341-354. doi: 10.1016/S0140-6736(20)32335-7. Epub 2021 May 27. PMID 34051884
- [Background] Abalos E, Cuesta C, Grosso AL, Chou D, Say L. Global and regional estimates of preeclampsia and eclampsia: a systematic review. Eur J Obstet Gynecol Reprod Biol. 2013 Sep;170(1):1-7. doi: 10.1016/j.ejogrb.2013.05.005. Epub 2013 Jun 7. PMID 23746796
- [Background] Cluver CA, Hiscock R, Decloedt EH, Hall DR, Schell S, Mol BW, Brownfoot F, Kaitu'u-Lino TJ, Walker SP, Tong S. Use of metformin to prolong gestation in preterm pre-eclampsia: randomised, double blind, placebo controlled trial. BMJ. 2021 Sep 22;374:n2103. doi: 10.1136/bmj.n2103. PMID 34551918
- [Background] Brownfoot FC, Hastie R, Hannan NJ, Cannon P, Tuohey L, Parry LJ, Senadheera S, Illanes SE, Kaitu'u-Lino TJ, Tong S. Metformin as a prevention and treatment for preeclampsia: effects on soluble fms-like tyrosine kinase 1 and soluble endoglin secretion and endothelial dysfunction. Am J Obstet Gynecol. 2016 Mar;214(3):356.e1-356.e15. doi: 10.1016/j.ajog.2015.12.019. Epub 2015 Dec 22. PMID 26721779
- [Background] Hu J, Zhang J, Zhu B. Protective effect of metformin on a rat model of lipopolysaccharide-induced preeclampsia. Fundam Clin Pharmacol. 2019 Dec;33(6):649-658. doi: 10.1111/fcp.12501. Epub 2019 Aug 13. PMID 31334867
- [Background] Wang F, Cao G, Yi W, Li L, Cao X. Effect of Metformin on a Preeclampsia-Like Mouse Model Induced by High-Fat Diet. Biomed Res Int. 2019 Dec 7;2019:6547019. doi: 10.1155/2019/6547019. eCollection 2019. PMID 31886236